CLINICAL TRIAL: NCT01281839
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled Study to Investigate the Efficacy, Safety and Tolerability of TMC435 vs Placebo as Part of a Treatment Regimen Including Peginterferon α-2a and Ribavirin in Hepatitis C, Genotype 1 Infected Subjects Who Relapsed After Previous Interferon-based Therapy
Brief Title: An Efficacy, Safety and Tolerability Study of TMC435 in Genotype 1 Hepatitis C-infected Patients Who Relapsed After Previous Therapy
Acronym: PROMISE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen R&D Ireland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR017371; TMC435HPC3007 (Other: Janssen R&D Ireland); 2010-021113-23 (EudraCT Number)
Record Dates: First submitted 2011-01-07; First posted 2011-01-24 (Estimated); Results first posted 2014-04-23 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-03

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; TMC435; HCV; Hep C; Genotype 1
MeSH Terms: conditions — Hepatitis C | interventions — Simeprevir; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TMC435 (Experimental): TMC435 150 mg capsule once daily for 12 weeks in addition to peginterferon alfa-2a and ribavirin for 24 or 48 weeks
  Interventions: Drug: TMC435; Drug: Peginterferon alpha-2a (PegIFN alpha-2a); Drug: Ribavirin (RBV)
- Placebo (Placebo Comparator): Placebo 150 mg capsule once daily for 12 weeks in addition to peginterferon alfa-2a and ribavirin for 48 weeks
  Interventions: Drug: Placebo; Drug: Peginterferon alpha-2a (PegIFN alpha-2a); Drug: Ribavirin (RBV)

INTERVENTIONS:
Drug: TMC435 — 150 mg capsule once daily for 12 weeks in addition to peginterferon alfa-2a and ribavirin for 24 or 48 weeks
  Arms: TMC435
Drug: Placebo — 150 mg capsule once daily for 12 weeks in addition to peginterferon alfa-2a and ribavirin for 48 weeks
  Arms: Placebo
Drug: Peginterferon alpha-2a (PegIFN alpha-2a) — One subcutaneous (under the skin) injection containing 0.5 mL solution with 180 mcg PegIFN alpha-2a once weekly for up to 48 weeks.
  Other Names: Pegasys
Drug: Ribavirin (RBV) — 200-mg tablets of RBV (body-weight adjusted dose) taken orally (by mouth) twice daily for up to 48 weeks.
  Other Names: Copegus

SUMMARY:
The purpose of this study is to investigate the effectiveness and safety of TMC435 compared with placebo in patients who are infected with genotype 1 hepatitis C virus who relapsed after previous interferon-based therapy. Patients will also receive peginterferon alfa-2a and ribavirin as part of their treatment.

DETAILED DESCRIPTION:
This is a randomized, double-blind (neither physician nor patients knows the name of the assigned drug), placebo-controlled study of TMC435 in patients who are infected with genotype 1 hepatitis C virus who relapsed after previous interferon-based therapy. Patients in this study will also receive two other drugs for their infection called peginterferon alfa-2a and ribavirin. The purpose of the study is to investigate if TMC435 is superior to placebo in reducing hepatitis C virus to an undetectable level 24 weeks after the end of treatment. For the first 12 weeks, patients will take TMC435 or placebo, plus peginterferon alfa-2a and ribavirin. For the next 12 weeks, patients will take peginterferon alfa-2a and ribavirin only. After that, some patients will continue to take peginterferon alfa-2a and ribavirin for up to 24 additional weeks. Other patients will stop taking peginterferon alfa-2a and ribavirin. The study doctor will inform each patient about how to take their study medication and when they should stop taking it. After a patient stops taking study medication, they will continue to come to the doctor's office for study visits until a total of 72 weeks after they enroll in the study. The total duration of the study is 78 weeks (including screening). Patients will be monitored for safety throughout the study. Study assessments at each study visit may include but are not limited to: blood and urine collection for testing, ECG assessments (a measurement of the electrical activity of your heart), patient questionnaires, and physical examinations TMC435 will be taken as an oral capsule of 150 mg once per day. Peginterferon (Pegasys ®) will be given as an injection of 180 µg once each week. Ribavirin (Copegus ®) will be taken as a tablet twice each day and the dose will depend on your body weight.

ELIGIBILITY:
Inclusion Criteria:

* Genotype 1 hepatitis C infection (confirmed at screening)
* Have previously received peginterferon-based therapy for at least 24 weeks with documented HCV RNA at last measurement and relapsed within 1 year of last taking medication
* Liver biopsy within 3 years before screening (or between the screening and baseline visit) showing chronic hepatitis C infection
* Must agree to use 2 forms of effective contraception throughout study (both males and females)

Exclusion Criteria:

* Infection with HIV or non-genotype 1 hepatitis C
* Liver disease not related to hepatitic C infection
* Hepatic decompensation
* Significant laboratory abnormalities or other active diseases
* Pregnant or planning to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 394 (Actual)
Dates: Start 2011-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen R&D Ireland Clinical Trial, Study Director — Janssen R&D Ireland
Locations (68):
- United States (11):
  - Bakersfield, California
  - Aurora, Colorado
  - Jacksonville, Florida
  - Orlando, Florida
  - Atlanta, Georgia
  - Crestview Hills, Kentucky
  - Saint Paul, Minnesota
  - Jackson, Mississippi
  - Germantown, Tennessee
  - Houston, Texas
  - San Antonio, Texas
- Australia (5):
  - Adelaide
  - Kingswood
  - Melbourne
  - Sydney
  - Woolloongabba
- Vienna, Austria
- Belgium (5):
  - Antwerp
  - Bruges
  - Brussels
  - Ghent
  - Leuven
- Canada (4):
  - Vancouver, British Columbia
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- France (7):
  - Créteil
  - Grenoble
  - Lyon
  - Nice
  - Paris
  - Rennes
  - Vandœuvre-lès-Nancy
- Germany (10):
  - Berlin
  - Düsseldorf
  - Frankfurt
  - Freiburg im Breisgau
  - Halle
  - Hamburg
  - Kiel
  - Leipzig
  - München
  - Würzburg
- New Zealand (3):
  - Auckland
  - Christchurch
  - Hamilton
- Poland (6):
  - Bialystok
  - Bydgoszcz
  - Czeladź
  - Kielce
  - Krakow
  - Warsaw
- Puerto Rico (2):
  - Ponce Pr
  - San Juan
- Russia (5):
  - Moscow
  - Saint Petersburg
  - Samara
  - Smolensk
  - Stavropol
- Spain (4):
  - Barcelona
  - Madrid
  - Seville
  - Valencia
- United Kingdom (5):
  - Birmingham
  - Derby
  - Glasgow
  - London
  - Plymouth

REFERENCES:
- [Derived] Lenz O, Verbinnen T, Fevery B, Tambuyzer L, Vijgen L, Peeters M, Buelens A, Ceulemans H, Beumont M, Picchio G, De Meyer S. Virology analyses of HCV isolates from genotype 1-infected patients treated with simeprevir plus peginterferon/ribavirin in Phase IIb/III studies. J Hepatol. 2015 May;62(5):1008-14. doi: 10.1016/j.jhep.2014.11.032. Epub 2014 Nov 28. PMID 25445400
- [Derived] Forns X, Lawitz E, Zeuzem S, Gane E, Bronowicki JP, Andreone P, Horban A, Brown A, Peeters M, Lenz O, Ouwerkerk-Mahadevan S, Scott J, De La Rosa G, Kalmeijer R, Sinha R, Beumont-Mauviel M. Simeprevir with peginterferon and ribavirin leads to high rates of SVR in patients with HCV genotype 1 who relapsed after previous therapy: a phase 3 trial. Gastroenterology. 2014 Jun;146(7):1669-79.e3. doi: 10.1053/j.gastro.2014.02.051. Epub 2014 Mar 3. PMID 24602923

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from 18 January 2011 to 4 February 2013. The study was conducted at 81 sites in 14 countries.
Pre-assignment Details: 394 participants were randomly allocated to the 2 treatment arms. 393 participants received at least 1 dose of study medication and were included in the intent-to-treat analysis set.
Groups:
- TMC435 150mg 12Wks PR24/48: Participants were given TMC435 150 mg once daily plus peginterferon alpha-2a (PegIFN alpha-2a) and ribavirin (RBV) for 12 Weeks (Wks) followed by PegIFN alpha-2a (P) and RBV (R) until Week 24 (PR24). Treatment was to be stopped at Week 24 for participants who achieved HCV RNA < 25 IU/mL detectable or undetectable at Week 4 and undetectable HCV RNA at Week 12. Other participants continued PR until Week 48 (PR48).
- PBO 12Wks PR48: Participants were given placebo (PBO) once daily plus peginterferon alpha-2a (PegIFN alpha-2a) and ribavirin (RBV) for 12 Weeks (Wks) followed by PegIFN alpha-2a (P) and RBV (R) until Week 48 (PR 48).
Period: Overall Study
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Started | 260 (Not including 1 participant was randomized to this group, but never received treatment.) | 133
Completed | 250 | 119
Not Completed | 10 | 14
Not completed — Lost to Follow-up | 6 | 3
Not completed — Withdrawal by Subject | 4 | 10
Not completed — Reason not specified | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48 | Total
Number analyzed (Participants) | 260 | 133 | 393
Age, Continuous [Median (Full Range); unit: years] | 52 [20 to 70] | 52 [21 to 71] | 52 [20 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 54 | 135
  Male | 179 | 79 | 258

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants Achieving a Sustained Virologic Response 12 Weeks After the Planned End of Treatment (SVR12)
Description: The table below shows the percentage of participants in each treatment group who achieved a SVR12, defined as the percentage of participants with undetectable plasma Hepatitis C virus ribonucleic acid 12 weeks after planned end of treatment.
Time Frame: Week 36 or Week 60
Population: The intent-to-treat population (defined as all participants who were randomized and received at least one dose of study medication) was used for all analyses.
Measure: Number; unit: Percentage of participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 260 | 133
Percentage of participants | 79.2 | 36.1
Statistical Analysis 1: Comparison: TMC435 150mg 12Wks PR24/48 vs PBO 12Wks PR48; Null hypothesis: There is no difference in proportions of SVR12 between the treatment groups; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Difference in proportions of SVR12 = 43.8, 95% CI 2-sided [34.6 to 53.0]

2. Secondary Outcome: The Percentage of Participants Achieving a Sustained Virologic Response at Week 72 (SVRW72)
Description: The table below shows the percentage of participants in each treatment group who achieved a SVRW72, defined as the percentage of participants with undetectable plasma Hepatitis C virus ribonucleic acid levels at end of treatment (EOT) and at Week 72.
Time Frame: Week 72
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 260 | 133
Percentage of Participants | 76.5 | 33.8
Statistical Analysis 1: Comparison: TMC435 150mg 12Wks PR24/48 vs PBO 12Wks PR48; Null hypothesis: There is no difference in proportions of SVR72 between the treatment groups; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Difference in proportions of SVR72 = 43.3, 95% CI 2-sided [34.1 to 52.5]

3. Secondary Outcome: The Percentage of Participants Who Achieved a Sustained Virologic Response 24 Weeks After the Planned End of Treatment (SVR24)
Description: The table below shows the percentage of participants in each treatment group who achieved a SVR24, defined as the percentage of participants with undetectable plasma Hepatitis C virus ribonucleic acid levels 24 weeks after planned end of treatment.
Time Frame: Week 48 or Week 72
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 260 | 133
Percentage of Participants | 77.3 | 33.8
Statistical Analysis 1: Comparison: TMC435 150mg 12Wks PR24/48 vs PBO 12Wks PR48; There is no difference in proportions of SVR24 between the treatment groups; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Difference in proportions of SVR24 = 44.1, 95% CI 2-sided [34.9 to 53.2]

4. Secondary Outcome: The Percentage of Participants Who Achieved a Sustained Virologic Response 4 Weeks After the Planned End of Treatment (SVR4)
Description: The table below shows the percentage of participants in each treatment group who achieved a SVR4, defined as the percentage of participants with undetectable plasma Hepatitis C virus ribonucleic acid levels 4 weeks after planned end of treatment.
Time Frame: Week 28 or Week 52
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 260 | 133
Percentage of Participants | 88.5 | 48.1
Statistical Analysis 1: Comparison: TMC435 150mg 12Wks PR24/48 vs PBO 12Wks PR48; There is no difference in proportions of SVR24 between the treatment groups; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Difference in proportions of SVR4 = 41.0, 95% CI 2-sided [32.1 to 49.9]

5. Secondary Outcome: Change From Baseline in log10 Hepatitis C Virus (HCV) Ribonucleic Acid (RNA)
Description: The table below shows change from baseline in log10 HCV RNA levels.
Time Frame: Day 3, Week 1, Week 4, Week 12, Week 24, and Week 48
Population: as for outcome 1
Measure: Mean (Standard Error); unit: log10 IU/mL
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 260 | 133
log10 IU/mL
  Day 3 | -3.537 (0.042) | -1.039 (0.072)
  Week 1 | -4.535 (0.040) | -1.099 (0.073)
  Week 4 | -5.295 (0.049) | -2.638 (0.125)
  Week 12 | -5.404 (0.049) | -4.476 (0.113)
  Week 24 | -5.449 (0.036) | -5.373 (0.070)
  Week 48 | -5.635 (0.212) | -5.473 (0.068)

6. Secondary Outcome: Actual Values of log10 Hepatitis C Virus (HCV) Ribonucleic Acid (RNA)
Description: The table below shows actual values of log10 HCV RNA levels. From Week 4 onwards, most participants in TMC 435 150mg 12Wks PR24/48 group had plasma HCV RNA levels below the limit of detection of the HCV RNA assay.
Time Frame: Day 3, Week 1, Week 4, Week 12, Week 24, and Week 48
Population: as for outcome 1
Measure: Mean (Standard Error); unit: log10 IU/mL
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 260 | 133
log10 IU/mL
  Day 3 | 2.884 (0.049) | 5.445 (0.084)
  Week 1 | 1.889 (0.041) | 5.376 (0.084)
  Week 4 | 1.128 (0.034) | 3.838 (0.130)
  Week 12 | 1.018 (0.034) | 2.005 (0.109)
  Week 24 | 0.956 (0.002) | 1.108 (0.042)
  Week 48 | 0.954 (0.000) | 0.995 (0.013)

7. Secondary Outcome: The Percentage of Participants With On-treatment Virologic Response at All Time Points
Description: The table below shows the percentage of participants with HCV ribonucleic acid (RNA plasma levels below the limit of detection (ie, <25 IU/mL undetectable), the percentage of participants with a HCV RNA plasma level below the limit of quantification (ie, less than [<] 25 IU/mL detectable or undetectable), the percentage of participants with plasma levels of HCV RNA <100 IU/mL, the percentage of participants with virologic responses of a greater than or equal to 2 log10 change from baseline in plasma levels of HCV RNA.
Time Frame: Day 3, Week 1, Week 2, Week 8, Week 16, Week 20, Week 28, Week 36, and Week 42
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 260 | 133
Percentage of Participants
  Day 3:<25 IU/mL undetectable | 0 | 0.8
  Week 1:<25 IU/mL undetectable | 3.9 | 0
  Week 2:<25 IU/mL undetectable | 28.3 | 0.8
  Week 8:<25 IU/mL undetectable | 95.7 | 15.0
  Week 16:<25 IU/mL | 98.4 | 47.4
  Week 20:<25 IU/mL | 99.6 | 65.5
  Week 28:<25 IU/mL | 88.9 | 84.5
  Week 36:<25 IU/mL | 90.0 | 91.9
  Week 42:<25 IU/mL | 100.0 | 91.7
  Day 3:<25 IU/mL undetectable/detectable | 3.1 | 0.8
  Week 1:<25 IU/mL undetectable/detectable | 35.9 | 0.8
  Week 2:<25 IU/mL undetectable/detectable | 82.6 | 1.5
  Week 8:<25 IU/mL undetectable/detectable | 98.0 | 27.6
  Week 16:<25 IU/mL undetectable/detectable | 100.0 | 77.6
  Week 20:<25 IU/mL undetectable/detectable | 99.6 | 89.4
  Week 28:<25 IU/mL undetectable/detectable | 100.0 | 100.0
  Week 36:<25 IU/mL undetectable/detectable | 90.0 | 99.0
  Week 42:<25 IU/mL undetectable/detectable | 100.0 | 97.9
  Day 3:<100 IU/mL | 9.1 | 0.8
  Week 1:<100 IU/mL | 62.2 | 0.8
  Week 2:<100 IU/mL | 92.2 | 2.3
  Week 8:<100 IU/mL | 98.0 | 37.0
  Week 16:<100 IU/mL | 100.0 | 84.5
  Week 20:<100 IU/mL | 99.6 | 93.8
  Week 28:<100 IU/mL | 100.0 | 100.0
  Week 36:<100 IU/mL | 90.0 | 100.0
  Week 42:<100 IU/mL | 100.0 | 100.0
  Day 3:> or = 2 log10 change from baseline | 97.6 | 14.1
  Week 1:> or = 2 log10 change from baseline | 99.6 | 13.7
  Week 2:> or = 2 log10 change from baseline | 99.6 | 35.4
  Week 8:> or = 2 log10 change from baseline | 98.4 | 87.4
  Week 16:> or = 2 log10 change from baseline | 100.0 | 100.0
  Week 20:> or = 2 log10 change from baseline | 100.0 | 100.0
  Week 28:> or = 2 log10 change from baseline | 100.0 | 100.0
  Week 36:> or = 2 log10 change from baseline | 100.0 | 100.0
  Week 42:> or = 2 log10 change from baseline | 100.0 | 100.0

8. Secondary Outcome: The Percentage of Participants Achieving a Rapid Virologic Response (RVR)
Description: The table below shows the percentage of participants in each treatment group who achieved a RVR, defined as having undetectable plasma Hepatitis C virus ribonucleic acid levels after receiving 4 weeks of treatment.
Time Frame: Week 4
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 260 | 133
Percentage of Participants | 77.2 | 3.1

9. Secondary Outcome: The Percentage of Participants Achieving a Early Virologic Response (EVR)
Description: The table below shows the percentage of participants who achieved an EVR, defined as having a change from baseline in plasma Hepatitis C virus ribonucleic acid of greater than or equal to 2 log10 at Week 12.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 260 | 133
Percentage of Participants | 98.8 | 95.2

10. Secondary Outcome: The Percentage of Participants Achieving a Complete Early Virologic Response (cEVR)
Description: The table below shows the percentage of participants in each treatment group who had a cEVR, defined as having undetectable plasma Hepatitis C Virus ribonucleic acid levels at Week 12.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 260 | 133
Percentage of Participants | 98.0 | 27.4

11. Secondary Outcome: The Percentage of Participants Achieving a Extended Rapid Virologic Response (eRVR)
Description: The table below shows the percentage of participants in each treatment group who had a eRVR, defined as having undetectable plasma Hepatitis C Virus ribonucleic acid levels at Week 4 and 12.
Time Frame: Week 4 and Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 260 | 133
Percentage of Participants | 77.6 | 1.6

12. Secondary Outcome: The Percentage of Participants With <1 log10 Decrease in Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) From Baseline at Week 4
Description: The table below shows the percentage of participants in each treatment group with <1 log10 HCV RNA decrease at Week 4.
Time Frame: Week 4
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 260 | 133
Percentage of Participants | 0.8 | 9.3

13. Secondary Outcome: Percentage of Participants With in Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Levels >1000 IU/mL at Week 4
Description: The table below shows the percentage of participants in each treatment group with HCV RNA levels >1000 IU/mL at Week 4.
Time Frame: Week 4
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 260 | 133
Percentage of Participants | 1.9 | 69.9

14. Secondary Outcome: The Percentage of Participants With Null Response
Description: The table below shows the percentage of participants with null response, defined as <2 log10 reduction in Hepatitis C virus ribonucleic acid at Week 12 compared to baseline.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 260 | 133
Percentage of Participants | 1.2 | 4.8

15. Secondary Outcome: The Percentage of Participants With Partial Response
Description: The table below shows the percentage of participants with partial response, defined as =>2 log10 reduction in Hepatitis C virus (HCV) ribonucleic acid (RNA) at Week 12 compared to baseline, but not achieving undetectable HCV RNA while on treatment.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 260 | 133
Percentage of Participants | 10.5 | 0

16. Secondary Outcome: The Percentage of Participants With Viral Breakthrough
Description: The table below shows the percentage of participants with viral breakthrough, defined as a confirmed increase of greater than 1 log10 IU/mL in plasma Hepatitis C virus (HCV) ribonucleic acid (RNA) level from the lowest level reached (ie, lowest value measured in between baseline and current value), or a confirmed plasma HCV RNA level of greater than 100 IU/mL in participants whose plasma HCV RNA had previously been below the limit of quantification (25 IU/mL detectable) or undetectable (<25 IU/mL undetectable).
Time Frame: Up to Week 48
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 260 | 133
Percentage of Participants | 0.0 | 2.3

17. Secondary Outcome: The Percentage of Participants With Viral Relapse
Description: The table below shows the percentage of participants with viral relapse, defined as having confirmed detectable plasma level of Hepatitis C virus (HCV) ribonucleic acid (RNA) during the follow-up period in participants with undetectable plasma HCV RNA (less than 25 IU/mL undetectable) at the end of treatment.
Time Frame: Up to Week 72
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 260 | 133
Percentage of Participants | 18.9 | 50.5

18. Secondary Outcome: The Percentage of Participants Who Completed All Study Treatment at Week 24 Because of the Treatment Duration Rule
Description: The table below shows the percentage of participants in the TMC435 treatment group who met the treatment duration rule (ie, having hepatitis C virus [HCV] ribonucleic acid [RNA] levels <25 IU/mL detectable or undetectable at Week 4 and undetectable HCV RNA levels at Week 12) and completed treatment with PegIFNα-2a and RBV for 24 weeks. Participants in the TMC435 treatment group not meeting RGT criteria and participants in the placebo group were treated with PegIFNα-2a and RBV treatment for 48 weeks.
Time Frame: Week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 260 | 133
Percentage of Participants | 90.0 | 0

19. Secondary Outcome: The Percentage of Participants With On-treatment Failure
Description: The table below shows percentage of participants with on-treatment failure defined as confirmed detectable Hepatitis C virus ribonucleic acid levels at actual end of treatment.
Time Frame: Week 48
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 260 | 133
Percentage of Participants | 3.1 | 27.1

20. Secondary Outcome: Time to Reach Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) <25 IU/mL Undetectable
Description: The table below shows mean time in days to reach HCV RNA levels <25 IU/mL undetectable or detectable.
Time Frame: Up to Week 48
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 260 | 133
Days | 28 [28 to 29] | 141 [113 to 167]

21. Secondary Outcome: Time to Reach Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) <25 IU/mL Undetectable or Detectable
Description: The table below shows mean time in days to reach HCV RNA levels <25 IU/mL undetectable or detectable.
Time Frame: Up to Week 48
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 260 | 133
Days | 14 [14 to 15] | 110 [85 to 113]

22. Secondary Outcome: Time to Reach Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) <100 IU/mL
Description: The table below shows mean time in days to reach HCV RNA levels <100 IU/mL.
Time Frame: Up to Week 48
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 260 | 133
Days | 8 [NA to NA] — 95% CI were not calculated because the number of censored values was very low (<5%) and the response occurred very rapidly in the responders (85% of the subjects had HCV RNA<100 IU/mL at Week 2). | 85 [83 to 85]

23. Secondary Outcome: Time to Reach Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) <1000 IU/mL
Description: The table below shows mean time in days to reach HCV RNA levels <1000 IU/mL.
Time Frame: Up to Week 48
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 260 | 133
Days | 4 [3 to 4] | 57 [57 to 58]

24. Secondary Outcome: The Percentage of Participants With Viral Breakthrough at Different Time Points
Description: The table below shows the percentage of participants at different time points with viral breakthrough, defined as a confirmed increase of greater than 1 log10 IU/mL in plasma HCV ribonucleic acid (RNA) level from the lowest level reached (ie, lowest value measured in between baseline and current value), or a confirmed plasma HCV RNA level of greater than 100 IU/mL in participants whose plasma HCV RNA had previously been below the limit of quantification (25 IU/mL detectable) or undetectable (<25 IU/mL undetectable).
Time Frame: Up to Week 48
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 260 | 133
Percentage of Participants
  =<12 weeks | 1.9 | 0.0
  >12-=<24 weeks | 0.0 | 0.0
  >24 weeks | 10.0 | 0.0

25. Secondary Outcome: Time From End-of-treatment to Viral Relapse
Description: The table below shows the mean number of days to viral relapse, defined as participants having confirmed detectable plasma level of Hepatitis C Virus (HCV) ribonucleic acid (RNA) during the follow-up period in participants with undetectable plasma HCV RNA (<25 IU/mL undetectable) at the end of treatment.
Time Frame: Up to Week 72
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Days
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 260 | 133
Days | 284.09 (6.56) | 115.22 (6.72)

26. Secondary Outcome: The Percentage of Participants With Normalization of Alanine Aminotransferase (ALT)
Description: The percentage of participants analyzed were those with baseline ALT values out of the normal range (ie, 156 of 260 participants in the TMC435 treatment group and 84 of 133 participants in the Placebo group had ALT values at baseline that were out of the normal range.). Normalization of ALT values means that ALT values out of the normal range returned to within the normal range.
Time Frame: Up to Week 48
Population: Participants with baseline ALT values out of normal range were used for this analysis from intent-to treat population (defined as all participants who were randomized and received at least one dose of study medication).
Measure: Number; unit: Percentage of Participants
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 156 | 84
Percentage of Participants | 69.9 | 69.0

27. Secondary Outcome: Median Time to Normalization of Alanine Aminotransferase (ALT) Levels
Description: The table below shows the median time to normalization of ALT levels.
Time Frame: Up to Week 48
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Number analyzed (Participants) | 260 | 133
Weeks | 7.86 [2.14 to 16.14] | 8.00 [4.14 to 15.86]

28. Secondary Outcome: Plasma Concentration of TMC435: Area Under the Plasma Concentration-time Curve From the Time of Administration to 24 Hours After Dosing (AUC24h)
Description: The table below shows mean (standard deviation) values of the area under the plasma concentration-time curve from time of administration to 24 hours (AUC 24hr) after dosing for TMC435. To calculate the mean AUC 24 for the study, AUC 24 hr values were derived for each participant at each visit and then the median of AUC value across visits for each participant was used to calculate the mean AUC 24 hr for the study.
Time Frame: From the time of administration up to 24 hours after dosing through Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | TMC435 150mg 12Wks PR24/48
Number analyzed (Participants) | 259
ng*h/mL | 60987 (67577.4) [2.14 to 16.14]

29. Secondary Outcome: Plasma Concentration of TMC435: Predose Plasma Concentration (C0h)
Description: The table below shows mean (standard deviation) of C0h values of TMC435. To calculate the mean C0h for the study, C0h values were derived for each participant at each visit and then the median of C0h values across visits for each participant was used to calculate the mean C0h for the study.
Time Frame: Before administration of TMC435 through Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | TMC435 150mg 12Wks PR24/48
Number analyzed (Participants) | 259
ng/mL | 2081 (2807.6) [2.14 to 16.14]

30. Secondary Outcome: Plasma Concentration of TMC435: Systemic Clearance (CL)
Description: The table below shows mean (standard deviation) of CL values of TMC435. To calculate the mean CL for the study, CL values were derived for each participant at each visit and then the median of CL values across visits for each participant was used to calculate the mean CL for the study.
Time Frame: From the time of administration through Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | TMC435 150mg 12Wks PR24/48
Number analyzed (Participants) | 259
L/h | 4.92 (3.438) [2.14 to 16.14]

ADVERSE EVENTS:
Time Frame: 72 weeks
Arm/Group | TMC435 150mg 12Wks PR24/48 | PBO 12Wks PR48
Serious Adverse Events (participants affected / at risk) | 14/260 | 11/133
Other Adverse Events (participants affected / at risk) | 245/260 | 123/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TMC435 150mg 12Wks PR24/48 (N=260) | PBO 12Wks PR48 (N=133)
Pneumonia (Infections and infestations) | 2 | 0
Appendicitis (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Arthritis infective (Infections and infestations) | 0 | 1
Bacterial prostatitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 1
Anaemia haemolytic autoimmune (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0
Guillain-Barre syndrome (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TMC435 150mg 12Wks PR24/48 (N=260) | PBO 12Wks PR48 (N=133)
Fatigue (General disorders) | 87 | 58
Influenza like illness (General disorders) | 78 | 27
Pyrexia (General disorders) | 63 | 30
Asthenia (General disorders) | 57 | 25
Injection site erythema (General disorders) | 21 | 9
Chills (General disorders) | 17 | 11
Pruritus (Skin and subcutaneous tissue disorders) | 72 | 37
Rash (Skin and subcutaneous tissue disorders) | 33 | 19
Alopecia (Skin and subcutaneous tissue disorders) | 26 | 17
Dry skin (Skin and subcutaneous tissue disorders) | 24 | 18
Eczema (Skin and subcutaneous tissue disorders) | 14 | 4
Erythema (Skin and subcutaneous tissue disorders) | 7 | 7
Headache (Nervous system disorders) | 87 | 48
Dizziness (Nervous system disorders) | 14 | 6
Dysgeusia (Nervous system disorders) | 12 | 7
Disturbance in attention (Nervous system disorders) | 10 | 7
Nausea (Gastrointestinal disorders) | 59 | 26
Diarrhoea (Gastrointestinal disorders) | 36 | 22
Vomiting (Gastrointestinal disorders) | 18 | 9
Abdominal pain upper (Gastrointestinal disorders) | 10 | 9
Abdominal pain (Gastrointestinal disorders) | 9 | 8
Insomnia (Psychiatric disorders) | 49 | 33
Mood altered (Psychiatric disorders) | 25 | 22
Depression (Psychiatric disorders) | 22 | 10
Sleep disorder (Psychiatric disorders) | 15 | 14
Depressed mood (Psychiatric disorders) | 10 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 34 | 21
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 26 | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 16 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 39 | 17
Arthralgia (Musculoskeletal and connective tissue disorders) | 26 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 8
Anaemia (Blood and lymphatic system disorders) | 40 | 24
Neutropenia (Blood and lymphatic system disorders) | 37 | 26
Decreased appetite (Metabolism and nutrition disorders) | 35 | 24
Nasopharyngitis (Infections and infestations) | 5 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days